CLINICAL TRIAL: NCT03709407
Title: "Effects of Different Manoeuvres of Manual Lymphatic Drainage in the Neck on Systems Nervous, Cardiovascular, Respiratory and Lymphatic in Healthy Subjects. Experimental Randomized Crossover Study"
Brief Title: "Effects of Manual Lymphatic Drainage in the Neck in Healthy Subjects. Experimental Randomized Crossover Study"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Angelo Rio, Principal Investigator, Universidad Europea de Madrid
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CIPI/029/17
Record Dates: First submitted 2018-10-10; First posted 2018-10-17 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2018-10

CONDITIONS: Blood Pressure; Nervous System Diseases, Sympathetic; Heart Rate Low; Lymphatic Diseases
MeSH Terms: conditions — Autonomic Nervous System Diseases; Bradycardia; Lymphatic Diseases | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- cervical stimuli (Experimental): Godoy´s maneuver with traction-sliding in supraclavicular fossa
  Interventions: Other: terminus; Other: Placebo; Other: Control group
- terminus (Experimental): Vodder´s maneuver with medial and anterior traction in supraclavicular fossa
  Interventions: Other: cervical stimuli; Other: Placebo; Other: Control group
- placebo (Sham Comparator): maneuver with sliding ON clavicular
  Interventions: Other: cervical stimuli; Other: terminus; Other: Control group
- Control group (No Intervention): only lying down

INTERVENTIONS:
Other: cervical stimuli — Manouvres Godoy
  Arms: placebo; terminus
Other: terminus — Manouvres Vodder
  Arms: cervical stimuli; placebo
Other: Placebo — placebo manouvre
  Arms: cervical stimuli; terminus
Other: Control group — lie down
  Arms: cervical stimuli; placebo; terminus

SUMMARY:
Drainage manoeuvres described in different Manual Lymphatic Drainage methods, suggest modificactions in vital signs, by changes at nervous system, that would involve modifications to heart rate, breathing rate, blood pressure, cardiac vascular level (arteries and lymphatics). In addition this hypothetical relaxing effect could be beneficial for other types of pathologies associated with the presence of stress, cardiac problems, respiratory pathology, muscle tension, muscle trigger points, etc. With this study investigators compare different manoeuvres in the neck area to observe the results in the participants regarding the basal state.

DETAILED DESCRIPTION:
Differentes drainage manoeuvres suggest changes at nervous system (sympathetic and parasympathetic nervous system) and other vital constants

ELIGIBILITY:
Inclusion Criteria:

* healthy men and women, physiotherapy students, to accept voluntarily participate and sign informed consent

Exclusion Criteria:

* systemic diseases, trauma history, neurological diseases, subjects with chronic pain, cardiovascular history of importance, depression, individuals who know the technique of MLD or that are under any medical treatment.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-03-19 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 8 times for 4 weeks
  Measured by validated tensiometer.

SECONDARY OUTCOMES:
range of movement | 8 times for 4 weeks
  Measured by validated goniometer CROM. 2 times for 4 weeks
pain pressure threshold | 8 times for 4 weeks
  Measured by validated analogical algometer
Respiratory rate | 8 times for 4 weeks
  Measured by observation
oxygen saturation | 8 times for 4 weeks
  Measured by validated pulseoximeter
Heart rate | 8 times for 4 weeks
  Measured by validated tensiometer and pulseoximeter

CONTACTS AND LOCATIONS:
Overall Officials: Angela Rio, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Angela, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided